CLINICAL TRIAL: NCT00723593
Title: Natural History and Pathophysiology of Gastrointestinal Graft Versus Host Disease
Brief Title: Natural History and Pathophysiology of Gastrointestinal Graft-versus-Host Disease
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080187; 08-DK-0187
Record Dates: First submitted 2008-07-25; First posted 2008-07-28 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2013-02-04

CONDITIONS: Graft-Versus-Host-Disease
Keywords: Graft-Versus-Host Disease; Gastrointestinal; Apoptotic Assay; Serum Proteomic Pattern Analysis; Mucosal Biopsy; Graft Versus Host Disease; GVHD
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will determine the best location to biopsy the gastrointestinal (GI) tract for early and accurate diagnosis of GI graft-versus-host-disease (GVHD). (A biopsy is the surgical removal of a small piece of tissue for examination under the microscope.) GVHD is a life-threatening complication of stem cell transplantation in which the donor s immune cells destroy the patient s healthy tissues. It most commonly affects the skin, liver and GI tract. This study will establish where to best biopsy tissue from the GI tract and study the tissue to try to explore how GI GVD occurs and how it may be possible to better diagnose and treat it.

Patients 18 years of age and older who have undergone or are who will undergo stem cell transplantation and who are at high risk for developing GI GVHD may be eligible for this study. Participants may enter the study before the transplant procedure or later if they develop GVHD symptoms.

Participants undergo the following tests and procedures:

I. Before starting conditioning chemotherapy or radiation therapy for the transplantation

* Medical history and physical examination
* Sigmoidoscopy (endoscopy of the lower part of the large intestine) and biopsies
* Blood draw
* Stool sample collection

II. Two to 3 weeks after conditioning regimen

* Sigmoidoscopy with biopsies
* Blood draw
* Stool sample collection

III. 30, 45, 60 and 90 days after transplantation

-Blood draw

IV. After completing the tests in part II and at the appearance of GI symptoms suspected to be due to GVHD

* Updated medical history and physical examination
* Esophagogastroduodenoscopy (endoscopy of the esophagus, stomach and upper small intestine)
* Colonoscopy (endoscopy of the entire part of the large intestine) with biopsies
* Blood draw
* Stool collection

V. Two weeks after starting therapy in patients diagnosed with GVHD

* Sigmoidoscopy with biopsies
* Blood draw
* Stool sample collection
* PET/CT scan in selected patients (nuclear medicine and x-ray imaging of the GI tract

DETAILED DESCRIPTION:
Graft-versus-host disease (GVHD) affects up to 70% of patients who undergo stem cell transplantation. GVHD is associated with significant morbidity and mortality, and commonly affects the skin, liver, and gastrointestinal (GI) system. Gastrointestinal (GI) manifestations of GVHD include anorexia, nausea, vomiting, abdominal pain, and diarrhea. In patients with GI GVHD, the extent of gut involvement and its relationship to underlying symptoms is unclear. Furthermore, diagnosis requires histologic evaluation that entails cumbersome invasive endoscopic procedures for tissue procurement. Histologic findings that support this diagnosis are nonspecific and have poor sensitivity and specificity. Treatment of GI GVHD is also nonspecific, and has many systemic side effects that account for a large portion of associated morbidity and mortality.

Such uncertainties regarding the diagnosis and treatment of GI GVHD stem from a lack of understanding of the pathophysiology of the disease. Cytokines produced by T lymphocytes, mononuclear phagocytes, and natural killer cells have been shown to play an integral role in the regulation of tissue damage. Human studies performed to date have examined peripheral blood cytokines, but results have been conflicting and with little clinical correlation. Current analysis of gut tissue has been limited mostly to animal subjects with little correlation to humans.

The primary objective of this study is to identify areas of the GI tract to be biopsied that would achieve the highest yield for the diagnosis of GI GVHD. This will be accomplished by performing esophagogastroduodenoscopy, colonoscopy, and ileoscopy in all post transplant patients with GI symptoms, suspected to be due to GVHD. Endoscopic biopsies will be evaluated by a single designated GI pathologist to make the diagnosis of GVHD. A novel application of a quantitative histological apoptotic assay will be evaluated in a blinded fashion for its diagnostic utility. A GVHD diagnostic yield rate for each area of the GI tract will be the primary outcome measure.

Other biopsies obtained at baseline, following the conditioning regimen as well as before and after therapy for GI GVHD will be used to achieve the secondary objective of understanding the immune response underlying GI GVHD. A comprehensive evaluation of the inflammatory milieu of gut tissues will be achieved using immunohistochemistry and flow cytometric immunophenotyping of mucosal mononuclear cells and microarray, qRT-PCR and ELISA of mucosal cytokines. Other secondary objectives include the evaluation of serum proteomic pattern analysis, serum citrulline, fecal calprotectin and 18F-FDG PET/CT for the noninvasive diagnosis of GI GVHD.

Better understanding of the pathophysiology of GI GVHD will allow us to develop more focused and effective diagnostic and therapeutic options that are less invasive and have fewer systemic side effects leading to reduced morbidity and mortality.

ELIGIBILITY:
* INCLUSION CRITERIA:

All patients 18 years or older who have undergone or plan to undergo any type of allogeneic bone marrow or peripheral stem cell transplant. (This will be coordinated with all different institutes at NIH to involve patients who participate in NIH affiliated protocols.)

EXCLUSION CRITERIA:

1. Patients who are under the age of 18 years.
2. Patients with a platelet count less than 30,000/mm(3).
3. Patients with an elevated prothrombin or partial thromboplastin time more than 1.5 times greater than the upper limit of normal or an absolute neutrophil count less than 500/mm(3) of blood or a history of a bleeding diathesis.
4. Women who are pregnant, as determined by laboratory evaluation performed according to the referring transplant protocol, or breast feeding.
5. Patients who are unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07-23; Study Completion 2013-02-04

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Wank, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)

REFERENCES:
- [Background] Cahn JY, Klein JP, Lee SJ, Milpied N, Blaise D, Antin JH, Leblond V, Ifrah N, Jouet JP, Loberiza F, Ringden O, Barrett AJ, Horowitz MM, Socie G; Societe Francaise de Greffe de Moelle et Therapie Cellulaire; Dana Farber Cancer Institute; International Bone Marrow Transplant Registry. Prospective evaluation of 2 acute graft-versus-host (GVHD) grading systems: a joint Societe Francaise de Greffe de Moelle et Therapie Cellulaire (SFGM-TC), Dana Farber Cancer Institute (DFCI), and International Bone Marrow Transplant Registry (IBMTR) prospective study. Blood. 2005 Aug 15;106(4):1495-500. doi: 10.1182/blood-2004-11-4557. Epub 2005 May 5. PMID 15878974
- [Background] Filipovich AH, Weisdorf D, Pavletic S, Socie G, Wingard JR, Lee SJ, Martin P, Chien J, Przepiorka D, Couriel D, Cowen EW, Dinndorf P, Farrell A, Hartzman R, Henslee-Downey J, Jacobsohn D, McDonald G, Mittleman B, Rizzo JD, Robinson M, Schubert M, Schultz K, Shulman H, Turner M, Vogelsang G, Flowers ME. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56. doi: 10.1016/j.bbmt.2005.09.004. PMID 16338616
- [Background] Martin PJ, McDonald GB, Sanders JE, Anasetti C, Appelbaum FR, Deeg HJ, Nash RA, Petersdorf EW, Hansen JA, Storb R. Increasingly frequent diagnosis of acute gastrointestinal graft-versus-host disease after allogeneic hematopoietic cell transplantation. Biol Blood Marrow Transplant. 2004 May;10(5):320-7. doi: 10.1016/j.bbmt.2003.12.304. PMID 15111931